CLINICAL TRIAL: NCT04256525
Title: The Efficacy and Safety of Prophylactic Anticoagulation for Catheter-related Thrombosis in Patients With Cancer and Implantable Venous Access Ports: a Prospective Multi-center Randomized Controlled Trial.
Brief Title: Prophylactic Anticoagulation for Catheter-related Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Research 2019-400
Record Dates: First submitted 2020-01-12; First posted 2020-02-05 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-01

CONDITIONS: Venous Thrombosis Due to Central Venous Access Device (Disorder); Prophylactic Anticoagulation; Patients With Tumor
Keywords: implantable venous access ports; Catheter Related thrombosis; thromboprophylaxis; anticoagulants; aspirin; low molecule heparin; rivaroxaban; cancer
MeSH Terms: conditions — Neoplasms | interventions — Rivaroxaban; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aspirin 100mg (Experimental)
  Interventions: Drug: Aspirin 100mg
- rivaroxaban 10mg (Experimental)
  Interventions: Drug: Rivaroxaban 10mg
- low molecule heparin (Experimental)
  Interventions: Drug: low molecule heparin
- Reference (No Intervention): mechanical prophylaxis

INTERVENTIONS:
Drug: Rivaroxaban 10mg — 10mg orally per day
  Arms: rivaroxaban 10mg
Drug: Aspirin 100mg — 100mg orally per day
  Arms: Aspirin 100mg
Drug: low molecule heparin — 0.4ml per day subcutaneous injection
  Arms: low molecule heparin

SUMMARY:
The main objective of this study is to compare the efficacy and safety of aspirin, low molecule heparin and rivaroxaban for preventing catheter-related thrombosis in middle-to-high-risk ambulatory patients with cancer and implantable venous access ports.

DETAILED DESCRIPTION:
Study Type: Interventional, randomized, parallel Assignment and no masking

Study Arms & Intervention: Drug 1: Aspirin, 100mg/day orally; Drug 2: rivaroxaban, 10mg/day orally; Drug 3: low molecule heparin, 4000IU(0.4ml)/day subcutaneous injection; Reference: mechanical prophylaxis.

Follow-up Period: 6 months. The trial visits occurred at time before each chemotherapy cycle. The following details should be included at each visit: Khorana score, height and weight, blood routine examination, coagulation function, stool-routine and occult blood test, renal and liver function, ultrasonography of both legs and neck.

Primary Outcome: The primary efficacy end point was the occurrence of thrombus in the vein at the puncture site or nearby. The primary was the occurrence of a major bleeding event as defined by the International Society on Thrombosis and Haemostasis (ISTH).

Secondary Outcome: The secondary efficacy end point was occurrence of occurrence of other thrombosis or embolism events like deep vein thrombosis or pulmonary embolism. The secondary safety endpoint was the occurrence of any clinically relevant non-major bleeding, minor bleeding and adverse events.

Population: patients with cancer and implantable venous access ports

Eligibility Criteria:

1. Age 18-75 years;
2. Patients with malignant tumors who received implantable drug delivery devices as intravenous access for systematic chemotherapy;
3. Eastern Cooperative Oncology Group (ECOG) class 0-1;
4. Expected to receive chemotherapy within 1 week of enrollment;
5. Expected survival of more than 6 months;
6. Ambulatory patients or outpatient chemotherapy patients whose intravenous chemotherapy less than 24 hours per hospital stay;
7. Khorana score 1-3 point.

Exclusion Criteria:

1. Patients with a history of allergies to low molecular weight heparin, rivaroxaban, aspirin or other non-steroidal anti-inflammatory drugs, especially those with asthma, neurovascular edema or shock;
2. Patients with bleeding risks: thrombocytopenia (platelet count < 50*109/L), clinically significant active bleeding, active gastric ulcer disease, severe arterial hypertension, history of previous stroke;
3. moderate to severe liver and kidney dysfunction;
4. pregnant or lactating women;
5. patients who are administered systemically with pyrrole-antimycotic agents (eg ketoconazole, itraconazole, voriconazole and posaconazole) or HIV protease inhibitors (eg ritonavir);
6. Patients taking methotrexate;
7. Patients with systemic use of non-steroidal anti-inflammatory drugs;
8. Patients who have had anticoagulant drugs for any other reason.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years;
2. patients with malignant tumors who received implantable drug delivery devices as intravenous access for systematic chemotherapy;
3. Eastern Cooperative Oncology Group (ECOG) class 0-1;
4. expected to receive chemotherapy within 1 week of enrollment;
5. expected survival of more than 6 months;
6. ambulatory patients or outpatient chemotherapy patients whose intravenous chemotherapy less than 24 hours per hospital stay;
7. Khorana score 1-3 point.

Exclusion Criteria:

1. patients with a history of allergies to low molecular weight heparin, rivaroxaban, aspirin or other non-steroidal anti-inflammatory drugs, especially those with asthma, neurovascular edema or shock;
2. patients with bleeding risks: thrombocytopenia (platelet count < 50*109/L), clinically significant active bleeding, active gastric ulcer disease, severe arterial hypertension, history of previous stroke;
3. moderate to severe liver and kidney dysfunction;
4. pregnant or lactating women;
5. patients who are administered systemically with pyrrole-antimycotic agents (eg ketoconazole, itraconazole, voriconazole and posaconazole) or HIV protease inhibitors (eg ritonavir);
6. patients taking methotrexate;
7. patients with systemic use of non-steroidal anti-inflammatory drugs;
8. patients who have had anticoagulant drugs for any other reason.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1640 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
occurrence of catheter-related thrombosis | from enrollment to the first time of occurrence of catheter-related thrombosis, up to 1 month after the completion of last chemotherapy cycle
  detect the occurrence of catheter-related thrombosis with ultrasound, venography if necessary
occurrence of major-bleeding event | from enrollment to the first time of occurrence of major-bleeding event, up to 1 month after the completion of last chemotherapy cycle
  define occurrence of major-bleeding event with ISTH standard

SECONDARY OUTCOMES:
occurrence of other thrombosis or embolism events except for catheter-related thrombosis | from enrollment to the first time of occurrence of other thrombosis or embolism events except for catheter-related thrombosis , up to 1 month after the completion of last chemotherapy cycle
  detect deep vein thrombosis with ultrasound for the lower extremity, , ultrasound for the upper extremity, pulmonary arteriography or venography if necessary
occurrence of clinically relevant non-major-bleeding, minor-bleeding or non-bleeding event | from enrollment to the first time of occurrence of events, up to 1 month after the completion of last chemotherapy cycle
  define occurrence of non-major-bleeding or minor-bleeding event with ISTH standard, evaluate the relevant adverse drug reaction with NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Doctor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (24):
- China (24):
  - the People's Hospital of Dongyang City, Dongyang, Zhejiang
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, the Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - the First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - the First People's Hospital of Xiaoshan District, Hangzhou, Hangzhou, Zhejiang
  - Women's Hospital of School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of TCM, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - the Central Hospital of Huzhou City, Huzhou, Zhejiang
  - the Second Affiliated Hospital of Jiaxing College, Jiaxing, Zhejiang
  - the Women's Hospital of Jiaxing City, Jiaxing, Zhejiang
  - the Central Hospital of Jinhua City, Jinhua, Zhejiang
  - the Central Hospital of Lishui City, Lishui, Zhejiang
  - the People's Hospital of Jinyun County, Lishui, Zhejiang
  - the People's Hospital of Lishui City, Lishui, Zhejiang
  - the Women's Hospital of Lishui City, Lishui, Zhejiang
  - the Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - the Huamei Hospital of Ningbo City, University of Chinese Academy of Sciences, Ningbo, Zhejiang
  - the People's Hospital of Yinzhou, Ningbo, Zhejiang
  - the Women's and Children's Hospital of Ningbo City, Ningbo, Zhejiang
  - the Affiliated Hospital of Shaoxing University, Shaoxing, Zhejiang
  - the First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - the Zhoushan Hospital of Zhejiang Province, Zhoushan, Zhejiang